CLINICAL TRIAL: NCT04467450
Title: Ultrasound Guided Botulinum Toxin Type A Injection of Subacromial-Subdeltoid Bursa in Hemiplegic Shoulder Pain: Comparative Study Versus Corticosteroid Injection
Brief Title: Ultrasound Guided Botulinum Toxin Type A Injection of Subacromial-Subdeltoid Bursa in Hemiplegic Shoulder Pain
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Eman Baraka, Assisstant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC6-5-2020
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Subacromial Bursitis; Subdeltoid Bursitis
Keywords: stroke; hemiplegia; botulinum toxin; musculoskeletal ultrasound
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Botulinum Toxins, Type A; methyl prednisolonate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox injection (Experimental): half of the hemiplegic patients will be injected by botulinum toxin A in the inflamed subacromial-subdeltoid bursa guided by musculoskeletal ultrasound
  Interventions: Drug: botulinum toxin type A
- methyl prednisolonate injection (Active Comparator): the other half of the hemiplegic patients will be injected by methylprednisolonate in the inflamed subacromial-subdeltoid bursa guided by musculoskeletal ultrasound
  Interventions: Drug: Methyl Prednisolonate

INTERVENTIONS:
Drug: botulinum toxin type A — ultrasound guided injection of the botulinum toxin type A in the inflamed subacromial subdeltoid bursa
  Other Names: botox 100 IU
  Arms: Botox injection
Drug: Methyl Prednisolonate — ultrasound guided injection of Methyl Prednisolonate in the inflamed subacromial subdeltoid bursa
  Other Names: Depomedrol 40mg /2ml
  Arms: methyl prednisolonate injection

SUMMARY:
Good shoulder function is a prerequisite for effective hand function, as well as for performing multiple tasks involving mobility, ambulation, and activities of daily living (ADL). A common sequela of stroke is hemiplegic shoulder pain, which can hamper functional recovery and subsequently lead to disability. Hemiplegic shoulder pain can begin as early as 2 weeks post stroke but typically occurs within 2-3 months post stroke.

DETAILED DESCRIPTION:
Subject and methods: Patients with clinical diagnosis of hemiparesis on the criteria of the World Health Organization (WHO, 2001) will be recruited from Benha university hospitals' outpatients and inpatients units of Rheumatology ,Rehabilitation and Physical medicine department The diagnosis of stroke was confirmed by the findings of either brain CT or MRI.

All patients should have localized severe shoulder pain of the paretic upper limb with or without limitation of shoulder range of motion (ROM) with the following inclusion criteria:

Hemiplegic shoulder pain (HSP) duration at least 3 months, pain score >3 on a pain visual analog scale (VAS) of 0 to 10 cm (0 no pain, 10 worst possible pain) at rest, and/or pain at movement score >5 on VAS during passive shoulder abduction, pain was not relieved by conventional treatment (common analgesics, such as paracetamol and non-steroidal anti-inflammatory drugs; slings; physical modalities such as transcutaneous electrical nerve stimulation of shoulder muscles or manual therapy). No significant spasticity in the upper shoulder joint, defined as Modified Ashworth Scale (MAS) score ≤2 , ultrasonographically diagnosed subacromial subdeltoid (SASD ) bursitis. previous shoulder steroid or botulinum toxin A injection in the affected side or known allergy for botulinum toxin.

Complete history will be addressed from all subjects emphasizing the age, sex, type of stroke (hemorrhagic, thrombotic) ,duration of the stroke, side of hemiplegia , duration of shoulder pain .Complete neurological and musculoskeletal examination .All patients will be examined by a single independent physiatrist.

Patients will be classified based on the type of the injected material into 2 categories: 18 patients will be injected by 20 IU botulinum Toxin A, ( BoNT/A) group and 18 patients will be injected by 40 mg methyl prednisolone (steroid group) The assessment of therapeutic effects will be performed at the start of the study, and in the 3rd and 10th weeks. Shoulder pain will quantified by VAS score at rest (night pain ) and during the day ( movement pain ) .

The physiatrist who will carry out the initial assessment and will perform the intra-articular injection will not participate in follow-up assessments.

Upper limb motor function was assessed sensorimotor function assessment for the upper extremity domain of the Fugl-Meyer Assessment (FMA-UE) .

Spasticity around the shoulder will be assessed by MAS. Physical disability and behavior related to activities of daily living will be assessed by Modified Barthel ADL index for stroke patients .

Subacromial subdeltoid bursitis(SASD) will be assessed in the paretic shoulder by high frequency probe SASD bursitis if there is thickness ≥ 2mm and / or effusion or both

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of hemiparesis caused by stroke diagnosed according to World Health Organization (WHO, 2001),
2. Shoulder pain for more than 3 months.
3. pain score >3 on a pain visual analog scale at rest.
4. pain score >5 on a pain visual analog scale during activity.
5. pain was not relieved by conventional treatment (common analgesics, and non-steroidal anti-inflammatory drugs, slings or physical modalities).
6. No significant spasticity in the upper shoulder joint, defined as Modified Ashworth Scale (MAS) score ≤2
7. Ultrasonographically diagnosed subacromial subdeltoid (SASD ) bursitis.

Exclusion Criteria :

1. history of shoulder pain or limited ROM before stroke.
2. previous trauma history affecting shoulder
3. shoulder subluxation
4. shoulder diseases ( osteoarthritis , rheumatoid arthritis , others )
5. other neurologic diseases
6. resistance greater than a MAS score 2
7. previous shoulder botulinum toxin or steroid injection in the affected side or known allergy for botulinum toxin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) for pain | One hour before the injection.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
visual analog scale (VAS) for pain | In the 1st follow up visit 2 weeks after the injection
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
visual analog scale (VAS) for pain | In the 2nd follow up visit 10 weeks after the injection .
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
The Modified Ashworth scale (MAS) | One hour before the injection
  measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity.[1] Scoring (taken from Bohannon and Smith, 1987):
  * 0: No increase in muscle tone
  * 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  * 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3: Considerable increase in muscle tone, passive movement difficult
  * 4: Affected part(s) rigid in flexion or extension
The Modified Ashworth scale (MAS) | In the 1st follow up visit 2 weeks after the injection
  measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity.[1] Scoring (taken from Bohannon and Smith, 1987):
  * 0: No increase in muscle tone
  * 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  * 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3: Considerable increase in muscle tone, passive movement difficult
  * 4: Affected part(s) rigid in flexion or extension
The Modified Ashworth scale (MAS) | In the 2nd follow up visit 10 weeks after the injection
  measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity.[1] Scoring (taken from Bohannon and Smith, 1987):
  * 0: No increase in muscle tone
  * 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  * 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3: Considerable increase in muscle tone, passive movement difficult
  * 4: Affected part(s) rigid in flexion or extension
Fugl-Meyer Assessment (FMA-UE) | One hour before the injection.
  The FM scale is a 226-point multi-item Likert-type scale developed as an evaluative measure of recovery from hemiplegic stroke. It is divided into 5 domains: motor function, sensory function, balance, joint range of motion, and joint pain. Each domain contains multiple items, each scored on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully).
  In our study we will assess only motor function domain of the upper limb excluding coordination testing and the total possible scale score for (FMA-UE) is 60.
Fugl-Meyer Assessment (FMA-UE) | In the 1st follow up visit 2 weeks after the injection
  The FM scale is a 226-point multi-item Likert-type scale developed as an evaluative measure of recovery from hemiplegic stroke. It is divided into 5 domains: motor function, sensory function, balance, joint range of motion, and joint pain. Each domain contains multiple items, each scored on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully).
  In our study we will assess only motor function domain of the upper limb excluding coordination testing and the total possible scale score for (FMA-UE) is 60.
Fugl-Meyer Assessment (FMA-UE) | In the 2nd follow up visit 10 weeks after the injection
  The FM scale is a 226-point multi-item Likert-type scale developed as an evaluative measure of recovery from hemiplegic stroke. It is divided into 5 domains: motor function, sensory function, balance, joint range of motion, and joint pain. Each domain contains multiple items, each scored on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully).
  In our study we will assess only motor function domain of the upper limb excluding coordination testing and the total possible scale score for (FMA-UE) is 60.
Modified Barthel ADL index* | One hour before the injection.
  Measure of physical disability used widely to assess behaviour relating to activities of daily living for stroke patients or patients with other disabling conditions. It measures what patients do in practice. Assessment is made by anyone who knows the patient well.
  Total score of 20 Score <15 - usually represents moderate disability <10- usually represents severe disability.
Modified Barthel ADL index* | In the 1st follow up visit 2 weeks after the injection
  Measure of physical disability used widely to assess behaviour relating to activities of daily living for stroke patients or patients with other disabling conditions. It measures what patients do in practice. Assessment is made by anyone who knows the patient well.
  Total score of 20 Score <15 - usually represents moderate disability <10- usually represents severe disability.
Modified Barthel ADL index* | In the 2nd follow up visit 10 weeks after the injection
  Measure of physical disability used widely to assess behaviour relating to activities of daily living for stroke patients or patients with other disabling conditions. It measures what patients do in practice. Assessment is made by anyone who knows the patient well.
  Total score of 20 Score <15 - usually represents moderate disability <10- usually represents severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Baraka, MD, Principal Investigator — Assisstant Profesoor
Locations (1):
- Eman, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee JH, Lee SH, Song SH. Clinical effectiveness of botulinum toxin type B in the treatment of subacromial bursitis or shoulder impingement syndrome. Clin J Pain. 2011 Jul-Aug;27(6):523-8. doi: 10.1097/AJP.0b013e31820e1310. PMID 21368663